CLINICAL TRIAL: NCT02544672
Title: Function Benefits of a Myoelectric Elbow-Wrist-Hand Orthosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Myomo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 15-260
Record Dates: First submitted 2015-09-01; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Cerebrovascular Accidents
MeSH Terms: conditions — Stroke

ARMS (1):
- Myoelectric Elbow-Wrist-Hand Orthosis (Experimental)
  Interventions: Device: Myoelectric Elbow-Wrist-Hand orthosis

INTERVENTIONS:
Device: Myoelectric Elbow-Wrist-Hand orthosis — An arm orthosis that uses myoelectric signals to control the level of mechanical assistance provided to a user's elbow and hand in order to overcome upper limb weakness or paralysis and achieve functional tasks.
  Other Names: MyoPro®

SUMMARY:
The objective of this study is to evaluate the functional benefits of a myoelectric Elbow-Wrist-Hand orthosis for persons with upper limb paralysis caused by a cerebrovascular accident (CVA).

DETAILED DESCRIPTION:
The objective of this study is to evaluate the functional gains provided by a myoelectric Elbow-Wrist-Hand orthosis for CVA patients with hemiparesis. The subjects will be fit with the device, provided general training in the operation of the EMG-controlled technology, and then guided through a series of standard clinical outcome measures used routinely as part of stroke rehabilitation medicine. The outcome measures employed in this study include the Fugl-Meyer assessment, the Box and Blocks test, and a battery of common functional tasks and activities. These outcome measures will allow the researchers to approximate the changes in the subjects' ability to successfully perform functional tasks with and without the MyoPro device.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years.
* Upper limb impairment caused by any stroke (CVA)
* Minimum of trace MMT (1/5) in Biceps and/or Triceps
* Full Passive range of motion in elbow, forearm, wrist, and hand
* Active shoulder flexion of at least 30 degrees of shoulder abduction of at least 20 degrees
* Score of at least 20 on the Mini Mental Status Examination.
* Ability to read and comprehend the English language.
* Ability to generate consistent, detectable EMG signal from the upper arm and forearm sensor sites with wrist in neutral or flexed positions.

Exclusion Criteria:

* Fixed upper limb contractures on affected side.
* Subjects with severe spasticity or tone (defined as 3 or more on the Modified Ashworth Scale).
* Inability to follow three step directions.
* Severe shoulder subluxation, pain or shoulder dislocation.
* Passive shoulder range of motion less than 45 degrees in flexion and abduction.
* Pain or hypersensitivity in the arm(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Upper Extremity (FMA-UE) | 2 hours
  Assessment of sensorimotor function for the upper extremities (arms)
  http://www.rehabmeasures.org/lists/rehabmeasures/dispform.aspx?ID=908
Modified Ashworth Scale | 2 hours
  Measurement of muscle spasticity due to nervous system injury or disease
  http://www.rehabmeasures.org/Lists/RehabMeasures/PrintView.aspx?ID=902
Box and Blocks Test | 2 hours
  An assessment of unilateral gross manual dexterity, measured by the number 1 inch cubes an individual can move over a barrier in a 60 second time period.
  http://www.rehabmeasures.org/Lists/RehabMeasures/DispForm.aspx?ID=917

CONTACTS AND LOCATIONS:
Locations (1):
- GRE Chardon, Chardon, Ohio, United States